CLINICAL TRIAL: NCT01583790
Title: A Prospective Trial for Laparoscopic Adjustable Gastric Banding in Morbidly Obese Patients: Report on Weight Loss, Metabolic Changes and Quality of Life
Brief Title: Factors Influencing the Positive Outcome of Bariatric Surgery for Morbidly Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Other Study IDs: AR-001-12
Record Dates: First submitted 2012-04-23; First posted 2012-04-24 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-03

CONDITIONS: Morbid Obesity; Diabetes; Hypertension
Keywords: Laparoscopic Sleeve Gastrectomy; Bariatric surgery; Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no group: laparoscopic sleeve gastrectomy

SUMMARY:
The purpose of this study is to report data with patients after bariatric surgery.

DETAILED DESCRIPTION:
In the period 2006-2012 the ICBS-Israeli Center for Bariatric Surgery in Assuta Hospital has performed about 1500 bariatric surgeries including Laparoscopic Adjustable Gastric Banding, Laparoscopic Sleeve Gastrectomy, Laparoscopic Roux en Y Gastric Bypass, and Duodenal switch. In addition, Pose and BPD procedures were performed.The ICBS team is comprised of a team of expert senior professionals in the obesity field, made up of the best bariatric surgeons, an expert endocrinologist who specializes in obesity and diabetes, a team of senior nutritionists and a supportive psychology team. During that period patients data were collected as part of the medical practice in the Center and included BMI, co-morbidities, weight loss programs the patients were involved in, pervious bariatric surgery and quality of life. During the entire 6 years of follow up data were collected which included weight loss, resolution of co-morbidity, changes in quality of life etc combined with training for healthy lifestyle.

The purpose of this retrospective study is to evaluate the key factors for surgery success that includes over 50% of original weight loss, resolution of co-morbidities. Factors that could affect surgical outcome such as age, repeated surgery, early side effects such as bleeding, leakage, thrombosis and lung emboli were recorded as well as later side effects such as herniation of the surgical area, production of gallbladder stones, vitamine deficiency and requirement of a revision surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients meeting established criteria set by the National Institutes of Health (NIH) for candidacy for bariatric surgery
* patients having a body mass index (BMI) of 35 with co-morbid conditions or BMI larger or equal 40 with or without co-morbid conditions,
* patients having a comorbidity that should be improved by the surgery
* Patients that are able to comprehend the risks and benefits and the surgical procedure
* patients having no glandular etiology for their obesity
* patients that have attempted to lose weight by conventional means
* patients that are willing to be observed over a long period of time

Exclusion Criteria:

* patients that can not obey one of the inclusion criteria

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes about 1500 patients, 70% female and 30% male. All patients that had bariatric surgery and were in the follow-up group for longer than one month will take part in the study. A special emphasis will be given to special population groups such as adolescents, old patients, patients undergoing revision surgery, and patients that required a additional type of surgery in conjunction with the bariatric surgery (e.g., gallbladder removal).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Weightloss of patients | At least one year

SECONDARY OUTCOMES:
Improvement of co-morbidities after surgery | At least one year
  Follow up visits were done at 1, 3, 6, 9, 12, 24, 36, 48 and 60 months after surgery. They included physical examinations, blood analysis and assessment of comorbidities in collaboration with attending family physician.

CONTACTS AND LOCATIONS:
Overall Officials: Asnat Raziel, MD, Principal Investigator — Medical Director, ICBS-Israeli Center for Bariatric Surgery
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel